CLINICAL TRIAL: NCT01630031
Title: Pulmonary Vein Isolation: Interest of Real-Time Contact Force Sensing During Radiofrequency Catheter Ablation for Paroxysmal Atrial Fibrillation
Brief Title: Contact Force Sensing and Pulmonary Vein Isolation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, JP Albenque, M.D., Clinique Pasteur
Other Study IDs: 1
Record Dates: First submitted 2012-06-23; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Paroxysmal Atrial Fibrillation; Catheter Ablation
Keywords: atrial fibrillation; paroxysmal; contact force; radiofrequency; catheter ablation; pulmonary vein isolation; recurrence; follow-up
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Use of the THERMOCOOL SF or EZ STEER THERMOCOOL Catheter, Biosense Webster, Inc.
- CF group: Use of THERMOCOOL SMARTTOUCH Catheter, Biosense Webster, Inc.

SUMMARY:
Introduction - Pulmonary vein isolation (PVI) is the cornerstone of paroxysmal atrial fibrillation (AF) ablation. Recurrences remain, however, not infrequent and are mainly due to PVs reconnection. In this setting, all procedural means able to improve the quality of tissue lesions are welcome.

Study Hypothesis - A continuous sensing of contact force (CF) during ablation, offered by a new catheter available on the market, was a valuable additional tool increasing the efficacy of the ablation procedure for PVI.

Methods - Prospective observational non-randomized monocentric study. Patients with paroxysmal AF receive PVI following standard ablation procedures (linear antral catheter ablation guided by CARTO 3 System, Biosense Webster, Inc.) using either a new irrigated RF ablation catheter that provides tip-to-tissue CF information (THERMOCOOL SMARTTOUCH Catheter, Biosense Webster, Inc.) (CF group), or a non-CF irrigated catheter (THERMOCOOL SF or EZ STEER THERMOCOOL Catheter, Biosense Webster, Inc.) (control group). Overall, 60 consecutive patients are enrolled in the study, with 30 patients in each group. All procedures is performed by the same experienced operator, not blinded to the catheter used. Except for CF information (with an objective of at least 10 g, associated to the most perpendicular vector obtainable), ablation procedures are carried out using identical approaches in both groups. Patients are discharged from hospital free of antiarrhythmic therapy. Patients are enrolled in a specific follow-up plan.

Primary Endpoints -(1) Proportion of PVI after exclusive anatomic approach, (2) Proportion of patients free of AF after 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal atrial fibrillation despite at least failure of one anti-arrhythmic drug
* Age 18-75 yrs
* First catheter ablation

Exclusion Criteria:

* Left ventricle ejection fraction at echocardiography <50%
* History of heart surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population included patients with paroxysmal atrial fibrillation who undergo a first catheter ablation procedure (pulmonary vein isolation).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of PVI after exclusive anatomic approach | Day 0
Proportion of patients free of AF after 12-month FU | One year

SECONDARY OUTCOMES:
Total time of fluoroscopy and radiation exposure | Day 0
Total time of RF application required for completed PVI | Day 0
Proportion of pericardial effusion at echocardiography | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Albenque, M.D., Principal Investigator — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, France

REFERENCES:
- [Derived] Marijon E, Fazaa S, Narayanan K, Guy-Moyat B, Bouzeman A, Providencia R, Treguer F, Combes N, Bortone A, Boveda S, Combes S, Albenque JP. Real-time contact force sensing for pulmonary vein isolation in the setting of paroxysmal atrial fibrillation: procedural and 1-year results. J Cardiovasc Electrophysiol. 2014 Feb;25(2):130-7. doi: 10.1111/jce.12303. Epub 2013 Nov 6. PMID 24433324